CLINICAL TRIAL: NCT07281846
Title: Transjugular Intrahepatic Portosystemic Shunt With or Without Branched-Chain Amino Acid Supplements in the Treatment of Patients With Cirrhotic Portal Hypertension Complicated by Sarcopenia: A Randomized Controlled Trial
Brief Title: TIPS With or Without BCAA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Collaborators: The First Affiliated Hospital of Zhengzhou University (Other); The First Affiliated Hospital of Henan University of Science and Technology (Other)
Responsible Party: Principal Investigator, Jiacheng Liu, Clinical Investigator, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TIPS-BCAA
Record Dates: First submitted 2025-12-02; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: BCAA; Cirrhosis; Portal Hypertension Related to Cirrhosis; Sarcopenia; Transjugular Intrahepatic Portosystemic Shunt
Keywords: Transjugular Intrahepatic Portosystemic Shunt; Sarcopenia; Portal Hypertension; Cirrhosis; BCAA
MeSH Terms: conditions — Fibrosis; Sarcopenia; Hypertension, Portal | interventions — Control Groups; Odorants

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study adopts a rigorous double-blind design to reduce bias, with specific implementations as follows: The placebo is prepared by an independent third-party institution not affiliated with the research team, and its appearance, odor, and packaging form are identical to those of the branched-chain amino acid (BCAA) supplement. It contains only inactive pharmaceutical excipients and has undergone safety evaluation, ensuring that the two cannot be distinguished by sensory characteristics; stratified block randomization is used for grouping: an independent third-party statistician generates a random allocation sequence via computer software (with gender and Child-Pugh classification as stratification factors and a dynamically adjusted block length of 4), and prepares sealed opaque envelopes to contain the grouping results. The envelopes are only opened by a research coordinator not involved in outcome assessment to confirm the grouping after the patient signs the informed consent form;
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BCAA Group (Experimental): The BCAA Group (experimental group) takes oral branched-chain amino acid (BCAA) supplements for 3 months starting after surgery.
  Interventions: Dietary Supplement: The BCAA Group (experimental group) takes oral branched-chain amino acid (BCAA) supplements for 3 months starting after TIPS.
- Non-BCAA Group (Placebo Comparator): The Placebo Group (control group) takes oral placebo for 3 months postoperatively-prepared by an independent third party, the placebo is identical to BCAA supplements in appearance, odor, and packaging to maintain blinding.
  Interventions: Dietary Supplement: The Placebo Group (control group) takes oral placebo for 3 months postoperatively-prepared by an independent third party, the placebo is identical to BCAA supplements in appearance, odor, and packagin

INTERVENTIONS:
Dietary Supplement: The BCAA Group (experimental group) takes oral branched-chain amino acid (BCAA) supplements for 3 months starting after TIPS. — This prospective randomized controlled trial (RCT) aims to compare changes in muscle mass and clinical outcomes between sarcopenic cirrhotic patients with portal hypertension and variceal bleeding who undergo transjugular intrahepatic portosystemic shunt (TIPS) plus branched-chain amino acid (BCAA) supplementation versus TIPS plus placebo. Eligible patients are aged 18-75 years, with cirrhosis, sarcopenia (defined by EASL guidelines: L3 skeletal muscle index [L3-SMI] <50 cm²/m² for males, <39 cm²/m² for females, measured via preoperative abdominal CT), and TIPS eligibility due to variceal bleeding or refractory ascites; exclusions include malignancies, severe cardiopulmonary insufficiency, Child-Pugh score >13, recurrent hepatic encephalopathy (HE), and prior use of nutrition supplements within 3 months. TIPS is standardized with 8mm covered Viatorr stents, intraoperative variceal embolization if needed, and a postoperative portal pressure gradient (PPG) target of <12 mmHg or ≥50% base
  Arms: BCAA Group
Dietary Supplement: The Placebo Group (control group) takes oral placebo for 3 months postoperatively-prepared by an independent third party, the placebo is identical to BCAA supplements in appearance, odor, and packagin — The Placebo Group (control group) takes oral placebo for 3 months postoperatively-prepared by an independent third party, the placebo is identical to BCAA supplements in appearance, odor, and packaging to maintain blinding.
  Arms: Non-BCAA Group

SUMMARY:
Cirrhosis is a major global cause of morbidity and mortality in chronic liver disease patients, accounting for 2.4% of global deaths in 2019. A 1990-2017 Global Burden of Disease study showed rising cirrhosis-related deaths, bringing heavy health and economic burdens. It often leads to portal hypertension and subsequent complications like ascites, gastroesophageal variceal bleeding (20% 6-week mortality), and hepatic encephalopathy (HE). Transjugular intrahepatic portosystemic shunt (TIPS) is an important treatment for variceal bleeding and refractory ascites per guidelines from EASL, AASLD, and the Chinese Medical Association.

Malnutrition affects 20% of compensated and over 50% of decompensated cirrhotic patients; sarcopenia (severe malnutrition) is linked to higher cirrhosis-related complications, impaired quality of life, survival, and poor prognosis in TIPS-treated patients. Thus, concurrent sarcopenia intervention during TIPS may improve outcomes.

Baveno VII, EASL, and AASLD guidelines recommend branched-chain amino acid (BCAA) and leucine-rich supplements for decompensated cirrhosis to ensure adequate nitrogen intake. RCT evidence shows BCAAs improve skeletal muscle index (SMI) in cirrhotic patients with sarcopenia and reduce HE risk, but evidence for TIPS-treated patients is lacking. This study aims to compare muscle mass changes and clinical prognosis between TIPS patients with sarcopenia, portal hypertension, and variceal bleeding who receive TIPS with or without BCAA supplements.

DETAILED DESCRIPTION:
Cirrhosis is a major cause of morbidity and mortality among patients with chronic liver disease worldwide. In 2019, cirrhosis accounted for 2.4% of global deaths. A Global Burden of Disease study (1990-2017) showed that the number of deaths caused by cirrhosis has been on the rise year by year since 1990, imposing a severe health and economic burden on many countries and peoples around the world. Cirrhosis is usually accompanied by the development of portal hypertension, which further leads to complications such as ascites, gastroesophageal variceal bleeding, and hepatic encephalopathy (HE). Among these, the mortality rate of gastroesophageal variceal bleeding reaches as high as 20% within 6 weeks of onset. Currently, according to guidelines issued by the European Association for the Study of the Liver (EASL), the American Association for the Study of Liver Diseases (AASLD), and the Chinese Medical Association, transjugular intrahepatic portosystemic shunt (TIPS) has become an important treatment for variceal bleeding and refractory ascites.

Malnutrition is a common complication of cirrhosis, affecting 20% of patients with compensated cirrhosis and more than 50% of those with decompensated cirrhosis. Sarcopenia is generally regarded as severe malnutrition, and its occurrence is often associated with a higher risk of cirrhosis-related complications (such as hepatic encephalopathy, ascites, and infections), which seriously impairs patients' quality of life and survival. Several studies have shown that sarcopenia is associated with poor prognosis in cirrhotic patients undergoing TIPS treatment. Therefore, concurrent intervention for sarcopenia during TIPS treatment may improve prognosis and thus enhance patient survival.

The Baveno VII guidelines point out that malnutrition increases the risk of poor prognosis in patients with cirrhosis and acute variceal bleeding, and oral nutrition should be initiated as soon as possible. Both the EASL Clinical Practice Guidelines on Nutrition in Chronic Liver Disease and the AASLD Practice Guidance on Malnutrition, Frailty, and Sarcopenia in Patients with Cirrhosis recommend the use of branched-chain amino acid (BCAA) supplements and leucine-rich amino acid supplements in patients with decompensated cirrhosis to achieve adequate nitrogen intake. An RCT study demonstrated that BCAA supplements can improve the skeletal muscle index (SMI) in cirrhotic patients with sarcopenia. Additionally, evidence suggests that BCAA supplements can significantly reduce the risk of hepatic encephalopathy (HE).

Therefore, BCAA supplements may serve as a routine nutritional supplement for cirrhotic patients undergoing TIPS treatment, but relevant evidence is currently lacking. This study aims to compare changes in muscle mass and clinical prognosis between cirrhotic patients with portal hypertension and variceal bleeding complicated by sarcopenia who receive TIPS with or without BCAA supplements, so as to verify our hypothesis.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 80 years old;
2. Diagnosed with cirrhosis complicated by sarcopenia;
3. Patients admitted due to variceal bleeding or refractory ascites who meet the indications for transjugular intrahepatic portosystemic shunt (TIPS).

Exclusion Criteria:

1. Hepatocellular carcinoma and/or other malignant tumors;
2. Severe cardiopulmonary insufficiency;
3. Child-Pugh score > 13 points;
4. Spontaneous recurrent hepatic encephalopathy (HE);
5. Large spontaneous portosystemic shunt;
6. Sepsis; spontaneous bacterial peritonitis (SBP);
7. Allergy to any component of the study nutritional supplement;
8. High-energy and high-protein diet or use of calcium supplements, vitamin D supplements, or protein/amino acid supplements within 3 months prior to the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2025-11-15 (Actual); Primary Completion 2027-11-15 (Estimated); Study Completion 2027-11-15 (Estimated)

PRIMARY OUTCOMES:
Differences in the sarcopenia reversal rate between the two groups (BCAA and Non-BCAA) | 1 year
  Sarcopenia is defined per the European Association for the Study of the Liver (EASL) clinical practice guidelines: the skeletal muscle index (SMI) is calculated as the ratio of the total cross-sectional area of all skeletal muscles at the third lumbar (L3) level (measured via abdominal CT, unit: cm²) to the square of height (unit: m²), with males having SMI < 50 cm²/m² and females < 39 cm²/m² diagnosed as sarcopenic. SMI is measured preoperatively and at 3 and 6 months post-TIPS to determine the reversal rate (proportion of patients no longer meeting sarcopenia criteria), and the difference in this rate between the two groups is compared to evaluate the effect of BCAA supplementation.
Differences in Short Physical Performance Battery (SPPB) scores between the two groups (BCAA and Non-BCAA) | 1 year
  The SPPB consists of three subtests: balance test, gait speed test, and Chair Stand Test. Each subtest is scored from 0 to 4 points, with a total score ranging from 0 to 12 points-higher scores indicate better physical fitness. The SPPB is assessed preoperatively and at 3 and 6 months post-TIPS to compare changes in physical performance between the BCAA and Non-BCAA groups, reflecting the effect of BCAA supplementation on functional capacity in cirrhotic patients with sarcopenia.

SECONDARY OUTCOMES:
The cumulative incidence of hepatic encephalopathy (HE) in the two groups (BCAA and Non-BCAA) | 1 year
  Hepatic encephalopathy (HE) is diagnosed and graded in accordance with the West-Haven criteria, with overt HE (OHE) defined as Grades II-IV. Data are collected during follow-up at 3 and 6 months after TIPS to compare whether branched-chain amino acid (BCAA) supplementation reduces the risk of HE compared with placebo. The Kaplan-Meier method is used to plot the cumulative incidence curves of HE in the two groups, and the Log-rank test is applied to compare the differences in the risk of HE occurrence between the two groups.
The cumulative incidence of death in the two groups (BCAA and Non-BCAA) | 1 year
  Death is defined as all-cause mortality occurring during the follow-up period after TIPS. Data on mortality events (including the time and cause of death) are collected through regular follow-up assessments at 3 and 6 months post-TIPS, as well as active follow-up via medical records and telephone inquiries for any unplanned hospitalizations or death reports. The aim is to compare whether branched-chain amino acid (BCAA) supplementation reduces the risk of death compared with placebo. The Kaplan-Meier method is used to plot the cumulative survival curves (and corresponding cumulative mortality curves) of the two groups, and the Log-rank test is applied to compare the differences in mortality risk between the two groups.
The cumulative incidence of Variceal Rebleeding in the two groups (BCAA and Non-BCAA) | 1 year
  Variceal rebleeding is diagnosed in accordance with the Baveno VII consensus criteria, defined as recurrent melena or hematemesis leading to any of the following: hospitalization, blood transfusion requirement, a decrease in hemoglobin of ≥3 g within 24 hours, or death within 6 weeks of the index bleeding event. Relevant data (including the time of rebleeding, clinical manifestations, and diagnostic evidence) are collected during scheduled follow-up at 3 and 6 months post-TIPS, as well as through emergency department and hospitalization records for acute bleeding episodes. The goal is to evaluate whether BCAA supplementation lowers the risk of variceal rebleeding compared with placebo. The Kaplan-Meier method is used to plot the cumulative incidence curves of variceal rebleeding in the two groups, and the Log-rank test is applied to compare the differences in rebleeding risk between the two groups.
The cumulative incidence of Shunt Dysfunction in the two groups (BCAA and Non-BCAA) | 1 year
  Shunt dysfunction is diagnosed based on the following criteria: color Doppler ultrasound detects a maximum shunt tract blood flow velocity ≤50 cm/s, ≥200 cm/s, or no blood flow signal; or recurrence of clinical symptoms (such as variceal rebleeding or refractory ascites) suggestive of shunt malfunction, which is further confirmed by transjugular portography showing >50% stenosis of the shunt tract. Data on shunt function are collected through color Doppler ultrasound examinations during follow-up at 3 and 6 months post-TIPS, as well as through portography for suspected cases. The purpose is to compare whether BCAA supplementation affects the risk of shunt dysfunction compared with placebo. The Kaplan-Meier method is used to plot the cumulative incidence curves of shunt dysfunction in the two groups, and the Log-rank test is applied to compare the differences in the risk of shunt dysfunction between the two groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, China

IPD SHARING:
Plan to Share IPD: Undecided